CLINICAL TRIAL: NCT03839030
Title: Development and Implementation of Mindfulness-Based Health Promotion Program for Educators (MBHP - Educa): Evaluation of Cognitive Functions and Epigenetic Modifications.
Brief Title: Mindfulness-Based Health Promotion Program for Educators (MBHP - Educa).
Acronym: Mindfulness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marcelo Demarzo, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Marcelo Demarzo, MD, PhD, Principal Investigator, Centro Mente Aberta de Mindfulness
Organization: Centro Mente Aberta de Mindfulness (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 92876418.2.0000.5505
Record Dates: First submitted 2018-10-15; First posted 2019-02-12 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Stress; Cognitive Impairment; Burnout Syndrome
MeSH Terms: conditions — Cognitive Dysfunction; Burnout, Psychological

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBHP-Educa (Experimental): Experimental: Intervention Group A novel Mindfulness-based Health Promotion program for Educators for active teachers will be employed. The intervention will be held once a week for 8-weeks, two-hour meetings (16.0-h total). Participants will be encouraged to meditate for 10-30 min/day via audio recording.
  Interventions: Other: MBHP-Educa
- Control Group (No Intervention): Control Group Teacher education as usual. These participants will participate in teacher training (Neuroscience for Education - Neuro Educa). The Neuro-Educa will be held once a week for 8-weeks, two-hour meetings (16.0-h total).

INTERVENTIONS:
Other: MBHP-Educa — This intervention is a meditative practice which the individuals will practice in their daily life following the MBHP-educa protocol
  Arms: MBHP-Educa

SUMMARY:
In the last few decades, the world has seen a significant increase in the occurrence of occupational diseases related to Burnout Syndrome (professional exhaustion) and stress in educators. These disorders affect mental health and teaching activity. In this way, they need to develop socio-emotional skills to cope with the psychosocial stressors related to the school environment. Currently, mindfulness-based therapies have been recommended to help educators acquire emotional self-control, and to improve self-esteem, metacognition, attention, resilience and affectivity, in addition to better the social skills needed in the school milieu. The main objective of the proposed research project is to elaborate a program of Mindfulness-Based Health Promotion - educators (MBHP - educa) to be applied to a population of Brazilian public school educators. The efficacy of the program will be evaluated by cognitive testing. Blood tests for the above-mentioned stress-related molecules will be performed. The goal of developing the MBHP - educa Program is to promote and ameliorate the health care of public school teachers. Developing such a research proposal will contribute to debate and implement public health policies focussed on promoting the health of public school teachers in Brazil.

DETAILED DESCRIPTION:
In the last few decades, the world has seen a significant increase in the occurrence of occupational diseases related to Burnout Syndrome (professional exhaustion) and stress in educators. These disorders affect mental health and teaching activity. In this way, they need to develop socio-emotional skills to cope with the psychosocial stressors related to the school environment. Currently, mindfulness-based therapies have been recommended to help educators acquire emotional self-control, and to improve self-esteem, metacognition, attention, resilience and affectivity, in addition to better the social skills needed in the school milieu. A few published studies indicate that mindfulness practices also reduce some inflammation- and stress- related molecules such as cortisol, receptor-interacting serine/threonine kinase 2 (RIPK2), cyclooxygenase 2 (COX2), interleukin 6 (IL-6), tumor necrosis factor-α (TNF-α) and epigenetic-regulation related histone deacetilases (HDAC). These indicator molecules can be measured in blood. The World Health Organisation (WHO-2013) recommends the worldwide implementation of strategies for the promotion of mental health, which are particularly aimed at preventing occupational diseases. The main objective of the proposed research project is to elaborate a program of Mindfulness-Based Health Promotion - educators (MBHP - educa) to be applied to a population of Brazilian public school educators. The efficacy of the program will be evaluated by cognitive testing. Blood tests for the above-mentioned stress-related molecules will be performed. The goal of developing the MBHP - educa Program is to promote and ameliorate the health care of public school teachers. Developing such a research proposal will contribute to debate and implement public health policies focussed on promoting the health of public school teachers in Brazil.

ELIGIBILITY:
Inclusion Criteria:

1)Brazilian male or female aged between 23 and 65 years and (2) currently working in the classroom

Exclusion Criteria:

(1) the presence of medical conditions or medications use that might affect inflammatory pathways; (2) report of an infectious condition in the last 15 days before collecting a blood sample; (3) active psychiatric and/or clinical comorbidities potentially life-threatening such as psychosis or suicidal ideation; and (4) had previously practiced or currently practicing meditation, yoga or Tai-Chi

Ages: 23 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2019-07-05 (Actual); Study Completion 2020-07-05 (Actual)

PRIMARY OUTCOMES:
World Health Organization Quality of Life-BREF (WHOQOL-BREF) | Pre-test, Post-test and follow-up (12 months)
  To evaluate quality of life through five subscales:
  physical domain - mean of responses psychological domain - mean of responses relationships domain - mean of responses environment domain - mean of responses quality of life and perception of life - mean of responses
  *each question response range one to five points Higher scores - Better Quality of Life
Pittsburgh Sleep Quality Index | Pre-test, Post-test and follow-up (12 months)
  To evaluate the Sleep Quality - sum of responses score
  *each questions have a specific conversion to range zero to six
  Higher scores - better sleep quality
Morningness-eveningness questionnaire - sum *Range 16 to 86 *higher scorer - more morningness type | Pre-test, Post-test and follow-up (12 months)
  To evaluate person's circadian rhythm (biological clock) (sum of all responses)

SECONDARY OUTCOMES:
Glutathione metabolism from blood samples | Pre-test, Post-test and follow-up (12 months)
  GSH plasma levels, Cysteine and homocisteine serum levels
Perceived Stress Scale (PSS-10) | Pre-test, Post-test and follow-up (12 months)
  to evaluate the level of subjectively noticed stress, composed of 10 items
Determination of cytokine levels in serum samples. | Pre-test, Post-test and follow-up (12 months)
  To evaluate the interleukin-8 (IL-8), interleukin-1β (IL-1β), interleukin-6 (IL-6), interleukin-10 (IL-10), tumor necrosis factor (TNF) e interleukin-12p70 (IL-12p70)
  *Concentration in micromol per liter. (mean and standard deviation, median and quartile per groups)
Connor-Davidson Resilience Rating Scale | Pre-test, Post-test and follow-up (12 months)
  The CD-RISC is a 25-item measure of resilience.
Positive and Negative Affect Schedule (PANAS) | Pre-test, Post-test and follow-up (12 months)
  To evaluate positive and negative Affect through two subscales:
  positive affect - sum negative affect - sum
  * each question range one to five
  * higher score - more frequent

OTHER OUTCOMES:
Five Facet Mindfulness Questionnaire (FFMQ) | Pre-test, Post-test and follow-up (12 months)
  To evaluate the mindfulness trace through five subscales:
  OBSERVING - mean DESCRIBING - mean NONJUDGE - mean NONREACT - mean ATC WITH AWARENESS - mean
  * each question range one to five
  * higher score - more mindful
Rey Auditory-Verbal Learning Test - RAVLT | Pre-test, Post-test and follow-up (12 months)
  To evaluate memory (number of word remember)
Stroop test | Pre-test, Post-test and follow-up (12 months)
  To evaluate attention and inhibitory behavior (number of errors and time)
Digit span test | Pre-test, Post-test and follow-up (12 months)
  To evaluate work memory (maximum lenght)
Trail Making Test - TMT | Pre-test, Post-test and follow-up (12 months)
  To evaluate attention (time to trail every letter or/and number)
Hospital Anxiety and Depression Scale (HAADS) | Pre-test, Post-test and follow-up (12 months)
  To evaluate anxiety and depression symptoms through two subscales:
  anxiety - sum depression - sum
  * each question range zero to four
  * higher score - more symptons
Burnout Clinical Subtypes Questionnaire - BCSQ-12 | Pre-test, Post-test and follow-up (12 months)
  To evaluate the burnout clinical subtypes through three subscales:
  Overload - mean, standard deviation and median Lack of development - mean, standard deviation and median Neglect - mean, standard deviation and median
  *each question response range one to seven points
  Higher scores - More Symptons of Burnout

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo MP Demarzo, PhD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Centro Mente Aberta de Mindfulness e Promoção de Saúde, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided